CLINICAL TRIAL: NCT02168374
Title: Biological and Physicomechanical Properties of Glass Ionomer Cements Associated With Chlorhexidine or Doxycycline
Brief Title: Properties of Glass Ionomer Cements Associated With Chlorhexidine or Doxycycline
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aline R F de Castilho (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor-Investigator, Aline R F de Castilho, Dr, University of Campinas, Brazil
Organization: University of Campinas, Brazil (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PGICACD; FAPESP (Other Grant/Funding Number: 2008/00359-0; 2008/02606-5)
Record Dates: First submitted 2014-06-03; First posted 2014-06-20 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Dental Caries
Keywords: Glass ionomer cement; Indirect pulp therapy
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Chlorhexidine - CHX (Experimental): Deciduous teeth were filled with GIC containing 1.25% chlorhexidine.
  Interventions: Other: Indirect pulp treatment
- Doxycycline - DOX (Experimental): Deciduous teeth were filled with GIC containing 4.5% doxycycline.
  Interventions: Other: Indirect pulp treatment
- Glass ionomer cement - GIC (Placebo Comparator): Deciduous teeth were filled with GIC without chlorhexidine or doxycycline.
  Interventions: Other: Indirect pulp treatment

INTERVENTIONS:
Other: Indirect pulp treatment — Carious dentine was sampled from the mesial portion of the cavity floor and the pulpal wall was entirely covered with one of the randomly selected materials: GIC containing 4.5% DOX; GIC containing 1.25% CHX or GIC as a control group. The antimicrobial concentrations were chosen based in the previous in vitro results obtained in this study. The cavities were then temporarily restored using a conventional GIC. Within 3 months after the initial treatment,the materials were carefully and completely removed, a new dentine sample was collected, and the teeth were then restored with a light-cured composite resin using a bonding system, after a new placement of the initial liner material.

SUMMARY:
This study assessed the clinical performance of a resin-modified glass ionomer cement containing different concentrations of chlorhexidine digluconate and doxycycline hyclate.

DETAILED DESCRIPTION:
This study aimed to evaluate the in vivo microbiologic action of the best concentration of chlorhexidine and doxycycline associated with the resin-modified glass ionomer cement applied on remaining dentine after indirect pulp treatment.

ELIGIBILITY:
Inclusion Criteria:

* an active deep carious lesion at the internal half of the dentine thickness of a primary molar that had not been previously restored and that involved the occlusal or occlusoproximal surface;
* the absence of signs of irreversible damage to the pulp
* the absence of radiolucencies at the interradicular or periapical region or thickening of the periodontal spaces, absence of internal and external root resorption, absence of calcification of the pulp tissue
* children presenting no systemic disease or those not using medications.

Exclusion Criteria:

* presence of signs of irreversible damage to the pulp
* children presenting systemic disease or those using medications.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2008-03; Primary Completion 2010-03 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Indirect Pulp Treatment using GIC associated with 1.25% CHX or 4.5% DOX. | up to 3 months
  Within 3 months after the initial treatment, the teeth were submitted to clinical and radiographic examination to determine signs and symptoms of pulp vitality.

SECONDARY OUTCOMES:
Indirect Pulp Treatment using GIC associated with 1.25% CHX or 4.5% DOX. | up to 3 months
  Dentine samples were collected at baseline and after 3 months of the treatment for microbiological evaluation (colony-forming unit - CFU).

CONTACTS AND LOCATIONS:
Overall Officials: Aline RF Castilho, PhD, Principal Investigator — Piracicaba Dental School, Unicamp

REFERENCES:
- [Result] de Castilho AR, Duque C, Negrini Tde C, Sacono NT, de Paula AB, de Souza Costa CA, Spolidorio DM, Puppin-Rontani RM. In vitro and in vivo investigation of the biological and mechanical behaviour of resin-modified glass-ionomer cement containing chlorhexidine. J Dent. 2013 Feb;41(2):155-63. doi: 10.1016/j.jdent.2012.10.014. Epub 2012 Oct 30. PMID 23123495